CLINICAL TRIAL: NCT06710795
Title: AFFIX: Evaluation of the performAnce and saFety of the MaxTack™ Motorized FIXation Device in Subjects Undergoing Repair of Ventral Hernia by Minimally Invasive Surgery
Brief Title: AFFIX: Post-market Study of MaxTack™ Motorized Fixation Device in Subjects Undergoing Ventral Hernia Repair
Acronym: AFFIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT23014
Record Dates: First submitted 2024-11-22; First posted 2024-11-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Masking Description: All subjects enrolled will receive the MaxTack™ Motorized Fixation Device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MaxTack™ Motorized Fixation Device (Experimental): Subjects treated with MaxTack™ Motorized Fixation Device when used for fixation of prosthetic material to soft tissue in minimally invasive ventral hernia repair
  Interventions: Device: MaxTack™ Motorized Fixation Device

INTERVENTIONS:
Device: MaxTack™ Motorized Fixation Device — All subjects enrolled will receive the MaxTack™ Motorized Fixation Device when used for fixation of prosthetic material to soft tissue in minimally invasive ventral hernia repair

SUMMARY:
Medtronic is sponsoring and funding the AFFIX study, a prospective, post-market, multicenter, nonrandomized, single-arm, interventional clinical study. The purpose of this study is to evaluate the performance and safety of the MaxTack™ Motorized Fixation Device when used for fixation of prosthetic material to soft tissue in minimally invasive ventral hernia repair procedures.

DETAILED DESCRIPTION:
A prospective, post-market, multicenter, nonrandomized, single-arm, interventional clinical study of the MaxTack™ Motorized Fixation Device when used for fixation of prosthetic material to soft tissue in minimally invasive ventral hernia repair procedures. Subjects will be followed in the short term (1 and 3 months) and long term (12 months) to evaluate safety and performance of the device.

The study is being conducted in two phases. Phase 1 will enroll approximately 33 subjects at up to 3 sites in the United States. Based on regulatory needs, Phase 2 may enroll additional subjects at approximately 10 US sites, for a total of up to 110 subjects across both phases.

ELIGIBILITY:
Preoperative Inclusion Criteria:

1. Subject has provided informed consent (IC)
2. Subject is 18 years of age or older at the time of consent
3. Subject is able and willing to comply with the study requirements and follow-up schedule
4. Subject is undergoing an elective, single-stage, primary or incisional ventral hernia repair
5. Subject is undergoing minimally invasive ventral hernia repair procedure using the MaxTack™ Motorized Fixation Device
6. Subject is undergoing minimally invasive ventral hernia repair procedure using a Medtronic (including Covidien) mesh that is intended to be used in compliance with the mesh Instructions for Use (IFU)
7. Subject is expected to meet the criteria for a class I wound (clean) as defined by Centers for Disease Control and Prevention (CDC) classification

Preoperative Exclusion Criteria:

1. Subject is undergoing an emergency surgery (e.g., lifesaving procedures performed where subject is in imminent danger of death, strangulated hernia, etc.)
2. Subject has history of 3 or more hernia repair procedures
3. Subject has existing mesh in the space where the physician needs to apply the new mesh to be fixated with the MaxTack™ Motorized Fixation Device
4. Subject is scheduled (or anticipated to be scheduled) for additional surgery, and subsequent surgery would jeopardize previous application of study treatment
5. Subject has history of allergic reactions to Poly (Glycolide-co-L-lActide) (PGLA)
6. Subject has history of allergic reactions to the components of the intended mesh
7. Subject has any systemic or local ongoing infection at the time of the surgery
8. Subject has a Body Mass Index (BMI) greater than 45 kg/m2
9. Subject has life expectancy in the opinion of the investigator, of less than 3 years at the time of enrollment
10. Subject is pregnant (as determined by standard site practices) or is planning to become pregnant during study duration period.
11. Subject has participated or will participate in an investigational drug or device research study that would interfere with the results of this study
12. Subject's participation in the study may jeopardize the safety or welfare of the subject, as determined by the investigator
13. Subject is already enrolled or was previously enrolled in this study

Intraoperative Exclusion Criteria:

1. Subject did not receive the MaxTack™ Motorized Fixation Device tacks to fixate the mesh
2. Subject did not receive a Medtronic (including Covidien) mesh
3. Inability to comply with the mesh IFU
4. Subject required more than a single piece of mesh
5. Subject has a surgical wound classified as Class II (clean-contaminated), Class III (contaminated) or Class IV (dirty/infected) as defined by the CDC classification
6. Subject with an American Society of Anesthesiologists (ASA) score of Class 4, 5, or 6
7. Inability to close the hernia defect
8. Subject's procedure required a multi-stage repair
9. Subject's minimally invasive procedure required to convert to open

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Surgical Site Occurrence (SSO) within 3 months following the MaxTack™ Motorized Fixation Device used for fixation in minimally invasive ventral hernia repair procedures. | 3-months
  The Phase 1 primary endpoint is the incidence of Surgical Site Occurrence (SSO) within 3 months following the use of the MaxTack™ Motorized Fixation Device for fixation in ventral hernia repair procedures. SSOs are considered Adverse Events (AEs) related to the study device, mesh, and/or study procedure and defined as Seroma, Hematoma, Surgical Site Infection (SSI), and bleeding at the tack implantation site.
  Note: Non-symptomatic seromas requiring no medical or surgical treatment are not reportable AEs. All symptomatic seromas as well as non-symptomatic seromas that require treatment, are considered reportable AEs.
Incidence of hernia recurrence within 3 months following the MaxTack™ Motorized Fixation Device used for fixation in minimally invasive ventral hernia repair procedures. | 3-months
  The Phase 2 primary endpoint is the incidence of hernia recurrence within 3 months following the use of MaxTack™ Motorized Fixation Device for fixation in minimally invasive ventral hernia repair procedures. Hernia recurrence is defined as a palpable fascial defect and/or a clinically manifested bulge, exacerbated by a Valsalva maneuver evaluated during a physical examination by the investigator and confirmed per site standard of care medical imaging, if necessary, at the respective clinical site. If a Valsalva maneuver is not conducted during physical examination, this must be reported as a protocol deviation.
  If standard of care imaging is done for hernia recurrence confirmation, the final decision to report a hernia recurrence will be based on the study investigator's assessment. Standard of care imaging may be done by a non-study, standard of care assessor, such as a radiologist.

SECONDARY OUTCOMES:
Incidence of Surgical Site Occurrence (SSO) | Discharge (post-surgery up to 1-month), 1-month, 12-months
  Incidence of Surgical Site Occurrence (SSO) which are the following AEs related to the study device, mesh, and / or study procedure and defined as seroma, hematoma, surgical site infection, bleeding at tack implantation site following the MaxTack™ Motorized Fixation Device used for fixation in minimally invasive ventral hernia repair procedures.
Incidence of SSO requiring Procedural Intervention (SSOPI) | Discharge (post-surgery up to 1-month), 1-month, 3-months, 12-months
  Incidence of SSO requiring Procedural Intervention (SSOPI) which are the following AEs related to the study device, mesh, and / or study procedure (seroma, hematoma, surgical site infection, bleeding at tack implantation site) following the MaxTack™ Motorized Fixation Device used for fixation in minimally invasive ventral hernia repair procedures.
Incidence of hernia recurrence | 1-month, 12-months
  Incidence of hernia recurrence following the MaxTack™ Motorized Fixation Device used for fixation in minimally invasive ventral hernia repair procedures. Hernia recurrence is defined as a palpable fascial defect and/or clinically manifested bulge, exacerbated by a Valsalva maneuver evaluated during a physical examination by the investigator and confirmed per site standard of care medical imaging, if necessary at the respective clinical site.
Incidence of hernia recurrences resulting in reoperation | 1-month, 3-months, 12-months
  Incidence of hernia recurrences resulting in reoperation, defined as an operative procedure performed with the specific goal of repairing the recurrent hernia.
Incidence of a MaxTack™ Motorized Fixation device deficiency (DD) | Operative Day (Day of Surgery)
  Incidence of MaxTack™ Motorized Fixation Device deficiencies (e.g., insufficient tack penetration, loose tacks, tack(s) migration, tacker issue battery etc.) on day of the index procedure.
Operative time for mesh fixation | Operative Day (Day of Surgery)
  Operative time for mesh fixation, defined as the time elapsed from the initiation of the mesh fixation process with MaxTack™ to its completion
Surgeon satisfaction | Operative Day (Day of Surgery)
  Surgeon satisfaction as assessed by Surgeon Satisfaction Questionnaire postoperatively.
Length of hospital stay | Discharge (post-surgery up to 1-month)
  Length of hospital stay after minimally invasive ventral hernia repair procedure where the MaxTack™ Motorized Fixation Device was used for fixation.
Change in Numeric Rating Scale (NRS) score | Screening compared to 1-month, 3-months, 12-months
  Change in subject-reported pain at the hernia site evaluated with Numeric Rating Scale (NRS) score from 0 to 10 at screening and compared to other timepoints. NRS is a unidimensional scale in which 11 numbers (between 0 and 10) are used to measure pain intensity. The patient is asked to choose the number that best reflects the pain intensity, with 0 = no pain and 10 = worst (unbearable) pain.
Change in Subject Quality of life (QoL) | Screening compared to 1-month, 3-months, 12-months
  Change in Subject Quality of life (QoL), as measured through the administration of the Hernia Quality of Life (HerQLes) questionnaire, evaluated at screening and compared to other timepoints. This is reported as a score from 0-100 with higher numbers indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Sachanandani, Study Director — Medtronic (Sponsor)
Locations (3):
- United States (3):
  - Cleveland Clinic - Weston Hospital, Weston, Florida
  - Cleveland Clinic - Ohio, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No